CLINICAL TRIAL: NCT02358811
Title: Evaluation of the Impact of Sleep Apnea on Cerebral Volumetry According to Age
Acronym: VOILAGE
Status: Terminated | Type: Observational
Why Stopped: change of Magnetic resonance imaging (MRI) research
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1308014; 2013-A00719-36 (Other: ANSM)
Record Dates: First submitted 2015-02-04; First posted 2015-02-09 (Estimated); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Obstructive Sleep Apnea (SAOS); Aging
Keywords: Obstructive Sleep Apnea; Voxel-Based Morphometry; Polysomnography; Magnetic resonance imaging
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Magnetic Resonance Imaging; Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Eldery SAOS+: Patients with severe obstructive sleep apnea (AHI>30) 70 years old and more
  Interventions: Device: Magnetic resonance imaging (MRI); Behavioral: Cognitive assessment
- Eldery SAOS-: People without obstructive sleep apnea (AHI<10) 70 years old and more
  Interventions: Device: Magnetic resonance imaging (MRI); Behavioral: Cognitive assessment
- Adult SAOS+: Patients with severe obstructive sleep apnea (AHI>30) 18 < Age < 55 years old
  Interventions: Device: Magnetic resonance imaging (MRI); Behavioral: Cognitive assessment
- Adult SAOS-: People without obstructive sleep apnea (AHI<10) 18 < Age < 55 years old
  Interventions: Device: Magnetic resonance imaging (MRI); Behavioral: Cognitive assessment

INTERVENTIONS:
Device: Magnetic resonance imaging (MRI) — The acquisition of the image will last 45 minutes with 6 sequences.
  * Before any examination, the manipulator will check the absence of contraindication to MRI.
  * During the fifth sequence, Gadolinium (Gadovist®) will be injected intravenously to the concentration 0.1 mmol / kg. For this, a venous catheter will be placed before the first sequence and then removed after the examination. This injection will be carried out according to the usual practice of MRI.
  * Throughout the examination, a physician will always be present.
Behavioral: Cognitive assessment — This cognitive assessment will include the following executive tests :
  * test of Stroop
  * left Trail Making Test A and B
  * verbal fluence test
  * test of memory of figures direct and inverse in order
  * completion of matrices
  * Paced Auditory Serial Addition Test (PASAT)

SUMMARY:
Sleep apnea is a common disease in the general population and more particularly in elderly subjects in whom prevalence can reach 30 % after 70 years old. In adults (<55 years old) cardiovascular consequences are well known and make sleep apnea treatment necessary. However elderly (>70 years old) apneic subjects are less symptomatic in terms of sleepiness, they usually present a lower index of respiratory events and cardiovascular consequences in this population are still discussed, driving some authors to consider sleep apnea in the elderly as a specific disease and making the need for a treatment questionable.

In this study the investigators will focus on the comparison between adult and elderly apneic subjects in terms of cognitive and cardiovascular consequences. Adult apneic patients suffer from a decrease of cognitive performance as well as grey matter local atrophy, particularly in the hippocampus and in the frontal lobes. According to fewer studies, white matter can also be affected by a demyelinisation process. These structural modifications are sometimes associated with disorders of executive and memory functions. In the elderly, no clear association can be drawn between cognitive decline and sleep apnea. Moreover, to our knowledge, the cerebral state of elderly symptomatic apneic subjects has mostly not be investigated.

DETAILED DESCRIPTION:
The goal of this project is to evaluate the impact of sleep apnea on the brain according to age. Our hypothesis is that adult apneic subjects would present local cerebral modification in the areas implied in cognition and memory, such as the hippocampus or the frontal areas, whereas elderly patients would present focal affects related to a deficit in the ventilatory and autonomic control without any major cognitive consequences.

Understanding the consequences of sleep apnea according to age could permit to refine the indications of sleep apnea treatment, mainly in elderly patients.

ELIGIBILITY:
Inclusion Criteria for patients:

* 18-55 or more than 70 years old
* SAOS (AHI>30) never treated before
* consent form signed

Inclusion Criteria for subjects:

* 18-55 or more than 70 years old
* No SAOS (AHI<10)
* consent form signed

Exclusion Criteria (subjects and patients) :

* Contraindication in the practice of MRI: pacemaker, metallic cardiac valve, intra-ocular metal part
* Contraindication in the injection of Gadolinium (allergy during a previous radiological examination).
* Type 1 or 2 diabetes
* History of cerebrovascular accident, myocardial infarction, congestive heart failure
* Chronic and/or severe renal insufficiency
* Chronic respiratory failure
* Neurological pathology
* Central origin sleep apnea (AHIcentral > 15)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects without SAOS and Patients with SAOS
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Level of grey of each of the voxels of the cerebral grey matter | During the MRI procedure
  We will use a technique widely used in neuroimage : the voxel-based morphometry (VBM) which allows a precise comparison by assessing local subtle differences at a voxel level (a voxel being a 3D-pixel).

SECONDARY OUTCOMES:
Level of grey of each of the voxels of the cerebral white matter | During the MRI procedure
  We will use a technique widely used in neuroimage : the voxel-based morphometry (VBM) which allows a precise comparison by assessing local subtle differences at a voxel level (a voxel being a 3D-pixel).
Cognitive score | At the inclusion
  It is the sum of the scores of the following tests :
  * test of Stroop
  * left Trail Making Test A and B
  * verbal fluence test
  * test of memory of figures direct and inverse in order
  * completion of matrices
  * Paced Auditory Serial Addition Test (PASAT)
Dosage of the markers of the inflammation | At the inclusion
  The blood markers of the inflammation are : C reactive protein (CRP US), Il1β, Il6, Il10, Tumor Necrosis Factor(TNFα) et Mitochondrial Pyruvate Carrier 1 (MPC1)

CONTACTS AND LOCATIONS:
Overall Officials: Frederic ROCHE, MD-PhD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No